CLINICAL TRIAL: NCT06524271
Title: Effect of Fermented Soybean (FSB) Supplementation on Gas-troesophageal Reflux Disease (GERD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NATTOME SDN BHD (Other)
Collaborators: UCSI University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nat0001
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Gastro Esophageal Reflux
Keywords: Gastroesophageal Reflux Disease (GERD); Reflux Disease Questionnaire (RDQ); inflammatory markers; Quality of Life in Reflux and Dyspepsia (QOLRAD)
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Same appearance of the supplements given. Identity of participant was masked during examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented soybean supplementation (Experimental): The intervention supplement composed of Lactobacillus delbrueckii FSB, hydrogen-ated palm kernel oil, sodium caseinate, isolated soy protein, brown rice, inulin, digestive enzymes blend (lactase, protease, cellulase, lipase, amylase, pectinase, papain, and bromelain), galacto-oligosaccharides (GOS), and Bifidobacterium longum, powder form packaged in individual sachets (NattomeTM, Nattome, Kuala Lumpur, Malaysia). The dosage of FSB in each sachet was 1g.
  Interventions: Dietary Supplement: Fermented Soybean
- Placebo control (Placebo Comparator): The placebo supplement had the exact composition of ingredients but excluding FSB.
  Interventions: Dietary Supplement: Supplement without fermented soybean

INTERVENTIONS:
Dietary Supplement: Fermented Soybean — Same as described earlier
  Other Names: Nattome
  Arms: Fermented soybean supplementation
Dietary Supplement: Supplement without fermented soybean — Same as described earlier
  Arms: Placebo control

SUMMARY:
Gastroesophageal reflux disease (GERD) is a prevalent chronic condition affecting the well-being of both adults and children in general medical practice. Research on the effects of fermented soy-bean (FSB) supplementation in managing GERD is relatively new, with limited studies available. Existing research often lacks sufficient dosing regimens and study durations to differentiate be-tween transient placebo effects and sustained benefits. In this study, the beneficial effects of FSB supplementation were investigated in 50 voluntary participants. Participants were required to take 1g of FSB supplement once daily for twelve weeks. GERD symptoms were evaluated using the Reflux Disease Questionnaire (RDQ), while inflammatory markers, including interleukin-4 (IL-4), interleukin-6 (IL-6), and interleukin-8 (IL-8), were measured to assess inflammation. The Quality of Life in Reflux and Dyspepsia (QOLRAD) questionnaire was used to evaluate partici-pants' quality of life. Results indicated that FSB supplementation significantly (P<0.05) alleviated heartburn and regurgitation symptoms and reduced levels of IL-4, IL-6, and IL-8, indicating a notable anti-inflammatory effect. Additionally, significant (P<0.05) improvements were observed in QOLRAD scores, particularly in vitality, emotional distress, and physical/social functioning. Collectively, our findings support the use of FSB as an adjuvant approach in managing GERD, with notable improvements in patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

(1) experienced heartburn, acid reflux, regurgitation, or non-cardiac chest pain within the past three months; (2) aged 18 years or older; (3) demonstrated the ability to comprehend the study protocol and information provided by the investigators; and (4) provided in-formed consent.

Exclusion Criteria:

1) use of medications related to GERD, such as acid inhibitors, antacids, prokinetics, gastric mucosal protectors, herbs, probiotics, or related preparations within the past two weeks; (2) a history of gastro-esophageal or duodenal surgery; (3) diagnosis of peptic ulcer, gastrointestinal bleeding, esophageal or gastric varices, or upper GI malignancies confirmed by endoscopy at tertiary hospitals; and (4) pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Reflux Disease Questionnaire (RDQ) | 4 weeks
  The RDQ assessed six symptoms across three domains (heartburn, regurgitation, and upper abdominal pain) using a 6-point Likert scale to measure frequency and severity over the preceding weeks
Quality of Life in Reflux and Dyspepsia (QOLRAD) | 4 weeks
  This questionnaire comprised 25 questions in five subdomains: emotional distress (questions 12, 14, 15, 17, 19, and 22), sleeping disorders (questions 8, 10, 11, 18, and 21), eating/drinking disorders (questions 3, 5, 9, 13, 16, and 20), physical/social function (questions 2, 6, 23, 24, and 25) and vitality (questions 1, 4, and 7). Participants rated each question on a 7-point Likert scale.
Inflammatory Markers | 4 weeks
  Three markers were assessed, namely IL-4, IL-6 and IL-8

CONTACTS AND LOCATIONS:
Locations (1):
- UCSI University, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request. All of the individual participant data collected during the trial, after deidentification will be shared upon reasonable request. Additional docu-ments including study protocol, statistical analysis plan, informed consent form and clinical study report will also be made available. The data will be available immediately following pub-lication with no end date. Data will be shared with anyone who wishes to access with reasonable request. The data can be used for any types of analyses.

REFERENCES:
- [Background] Shaw M, Dent J, Beebe T, Junghard O, Wiklund I, Lind T, Johnsson F. The Reflux Disease Questionnaire: a measure for assessment of treatment response in clinical trials. Health Qual Life Outcomes. 2008 Apr 30;6:31. doi: 10.1186/1477-7525-6-31. PMID 18447946
- [Background] Wiklund IK, Junghard O, Grace E, Talley NJ, Kamm M, Veldhuyzen van Zanten S, Pare P, Chiba N, Leddin DS, Bigard MA, Colin R, Schoenfeld P. Quality of Life in Reflux and Dyspepsia patients. Psychometric documentation of a new disease-specific questionnaire (QOLRAD). Eur J Surg Suppl. 1998;(583):41-9. PMID 10027672